CLINICAL TRIAL: NCT02173171
Title: A Registry Study to Evaluate the Survival and Long-Term Safety of Subjects Who Previously Received Talimogene Laherparepvec in Amgen or BioVEX-Sponsored Clinical Trials
Brief Title: Registry Study for Talimogene Laherparepvec
Status: Completed | Type: Observational
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Other Study IDs: 20120139
Record Dates: First submitted 2014-06-11; First posted 2014-06-24 (Estimated); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Any Tumor Type Eligible for Treatment With Talimogene Laherparepvec in Amgen or BioVEX-sponsored Clinical Trial
Keywords: Melanoma; talimogene laherparepvec
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Previously treated with T-VEC: Received at least 1 dose of talimogene laherparepvec on Amgen or BioVEX-sponsored clinical trial
  Interventions: Other: Information collection

INTERVENTIONS:
Other: Information collection — Q3M Information collection
  Other Names: Q3M Information collection

SUMMARY:
A Registry Study to Evaluate the Survival and Long-Term Safety of Subjects Who Previously Received Talimogene Laherparepvec in Amgen or BioVEX-Sponsored Clinical Trials

DETAILED DESCRIPTION:
A registry study is to evaluate the overall survival, use of subsequent anti-cancer therapy, and the long-term safety of subjects who have received at least one dose of talimogene laherparepvec on an Amgen or BioVEX-sponsored clinical trial for any tumor type. Follow-Up will occur every 3 months.

ELIGIBILITY:
Inclusion Criteria:

All subjects must provide informed consent prior to initiation of any study activities.

All subjects must have received at least one dose of talimogene laherparepvec on an Amgen or BioVEX-sponsored clinical trial for any tumor type and must have discontinued treatment and participation, including long-term follow-up (if applicable) in that trial.

Exclusion Criteria:

Subjects currently receiving talimogene laherparepvec in Amgen or BioVEX-sponsored clinical trial.

Subject currently participating, including for long-term follow-up (if applicable), in other Amgen-sponsored talimogene laherparepvec clinical trial.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who have received at least one dose of talimogene laherparepvec in an Amgen or BioVEX-sponsored clinical trial.
Sampling Method: Non-Probability Sample
Enrollment: 185 (Actual)
Dates: Start 2010-04-27 (Actual); Primary Completion 2021-09-23 (Actual); Study Completion 2021-09-23 (Actual)

PRIMARY OUTCOMES:
Talimogene Laherparepvec Related Adverse Events | 7 years
  Long-term safety of talimogene laherparepvec will be assessed by reporting of related adverse events every 3 months. Related serious adverse events will be reported within 24 hours following investigator's knowledge of the event.
Subject overall survival | 7 years
  Overall survival status will be reported every 3 months
Use of subsequent anti-cancer therapy | 7 years
  The use of subsequent anti-cancer therapy, for the tumor indication in the prior Amgen or BioVEX-sponsored clinical trial, including retreatment with marketed talimogene laherparepvec for approved indication in subjects previously enrolled in Amgen or BioVEX-sponsored talimogene laherparepvec clinical trials, will be monitored

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (59):
- United States (26):
  - University of South Alabama Mitchell Cancer Institute, Mobile, Alabama
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - St Joseph Heritage Healthcare, Santa Rosa, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - Florida Hospital Memorial Division, Daytona Beach, Florida
  - Baptist MD Anderson Cancer Center, Jacksonville, Florida
  - Mount Sinai Comprehensive Cancer Center, Miami Beach, Florida
  - H Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Oncology Specialists SC, Park Ridge, Illinois
  - Investigative Clinical Research of Indiana, LLC, Indianapolis, Indiana
  - Allina Health System dba Virginia Piper Cancer Institute, Minneapolis, Minnesota
  - Saint Louis University Hospital, St Louis, Missouri
  - Morristown Medical Center, Morristown, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - University of North Carolina Chapel Hill, Chapel Hill, North Carolina
  - Wake Forest Baptist Health Medical Center, Winston-Salem, North Carolina
  - Gabrail Cancer Center, LLC, Canton, Ohio
  - Providence Oncology and Hematology Care Eastside, Portland, Oregon
  - Greenville Health System Institute for Translational Oncology Research, Greenville, South Carolina
  - The West Clinic PC dba West Cancer Center, Germantown, Tennessee
  - Henry Joyce Cancer Center, Nashville, Tennessee
  - Mary Crowley Cancer Research, Dallas, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Intermountain Medical Center, Murray, Utah
  - University of Utah Huntsman Cancer Institute, Salt Lake City, Utah
  - Wheaton Franciscan Healthcare, Franklin, Wisconsin
- Austria (2):
  - Landeskrankenhaus Salzburg, Salzburg
  - Universitaetsklinikum Allgemeines Krankenhaus Wien, Vienna
- Canada (3):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - Princess Margaret Cancer Centre, Toronto, Ontario
- France (2):
  - Hopital Ambroise Pare, Boulogne-Billancourt
  - Centre Hospitalier Universitaire de Nantes, Hôpital Hôtel Dieu, Nantes
- Germany (2):
  - University Hospital, Heidelberg
  - Universitätsklinikum Tübingen, Tübingen
- Greece (3):
  - General Hospital of Athens Laiko, Athens
  - Metropolitan Hospital, Athens
  - Bioclinic of Thessaloniki, Thessaloniki
- Hungary (2):
  - Pecsi Tudomanyegyetem Klinikai Kozpont, Pécs
  - Szegedi Tudomanyegyetem Szent-Gyorgyi Albert Klinikai Kozpont Altalanos Orvostudomanyi Kar, Szeged
- Italy (3):
  - Azienda Socio Sanitaria Territoriale Papa Giovanni XXIII, Bergamo
  - IRCCS Istituto Europeo di Oncologia, Milan
  - Azienda Ospedaliera Universitaria Senese Policlinico Le Scotte, Siena
- Narodowy Instytut Onkologii im Marii Sklodowskiej-Curie - Panstwowy Instytut Badawczy, Warsaw, Poland
- Russia (2):
  - FSBI N N Blokhin Russian Oncology Research Center Ministry of Health of Russian Federation, Moscow
  - FSBI Scientific and Research Oncology Institute named after N N Petrov, Saint Petersburg
- Wilgers Oncology Centre, Pretoria, South Africa
- Yonsei University Health System Severance Hospital, Seoul, South Korea
- Spain (4):
  - Onkologikoa, Donostia / San Sebastian, Basque Country
  - Hospital Clinic i Provincial de Barcelona, Barcelona, Catalonia
  - Hospital General Universitario de Valencia, Valencia, Valencia
  - Hospital Universitario 12 de Octubre, Madrid
- Switzerland (4):
  - Kantonsspital Graubuenden, Chur
  - Hopitaux Universitaires de Geneve, Geneva
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - Universitaetsspital Zuerich, Zuerich Flughafen
- United Kingdom (3):
  - Guys and St Thomas Hospital, London
  - Royal Marsden Hospital, London
  - The Clatterbridge Cancer Centre NHS Foundation Trust, Metropolitan Borough of Wirral

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
  Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be
URL: https://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com